CLINICAL TRIAL: NCT05525468
Title: A Randomized, Double-blind, Vehicle-controlled, Parallel Group, Dose Escalation Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of TDM-180935 Following Topical Administration in Healthy Male Subjects
Brief Title: A Phase 1 Study of TDM-180935 Following Topical Administration in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Technoderma Medicines Inc. (Industry)
Collaborators: Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 239-13851-101
Record Dates: First submitted 2022-08-24; First posted 2022-09-01 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2022-08

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: A Randomized, Double-Blind, Vehicle-Controlled, Parallel Group, Dose Escalation Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of TDM-180935 Following Topical Administration in Healthy Male Subjects
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- SAD Cohorts 1-4 TDM-180935 topical ointment (Experimental): Single dose administration of TDM-180935 topic ointment, 0.25% or 0.5% or 1.0% or 2.0%
  Interventions: Drug: TDM-180935
- SAD placebo for TDM-180935 topical ointment (Placebo Comparator): Single dose administration of placebo for TDM-180935 topic ointment
  Interventions: Drug: Placebo
- MAD Cohorts 1-4 TDM-180935 topical ointment (Experimental): Multiple dose administration of TDM-180935 topic ointment, 0.25% or 0.5% or 1.0% or 2.0%
  Interventions: Drug: TDM-180935
- MAD placebo for TDM-180935 topical ointment (Placebo Comparator): Multiple dose administration of placebo for TDM-180935 topic ointment
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TDM-180935 — TDM-180935 topical ointment
  Arms: MAD Cohorts 1-4 TDM-180935 topical ointment; SAD Cohorts 1-4 TDM-180935 topical ointment
Drug: Placebo — Placebo for TDM-180935 topical ointment
  Arms: MAD placebo for TDM-180935 topical ointment; SAD placebo for TDM-180935 topical ointment

SUMMARY:
Multi-center, randomized, double-blind, vehicle-controlled, parallel group, dose escalation study of TDM-180935 following topical administration in healthy male subjects, 18 to 55 years old

DETAILED DESCRIPTION:
Protocol 239-13851-101 is a planned Phase 1 study entitled "A Randomized, Double-Blind, Vehicle-Controlled, Parallel Group, Dose Escalation Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of TDM-180935 Following Topical Administration in Healthy Male Subjects". Eligible subjects will be assigned to a sequential treatment cohort and randomized to each treatment group (active/placebo vs. placebo/placebo). Subject enrollment will continue into the next cohort after review of the dose safety from the previous dose cohort.

ELIGIBILITY:
Inclusion Criteria:

To enter the study, a subject must meet the following criteria:

1. Subject is a male, 18-55 years old at Visit1/Screening.
2. Subject has provided written informed consent.
3. Subject is willing and able to apply the IP(s) as directed, comply with study instructions (including avoiding direct sunlight exposure to the areas of IP application), and commit to all follow-up visits for the duration of the study.
4. Subject, in the investigator's opinion, is in good general health and free of any disease state or physical condition that might impair evaluation or exposes the subject to an unacceptable risk by study participation.
5. Subject has normal renal and hepatic function as determined by the Visit 1/Screening laboratory results in the opinion of the investigator.
6. Subject is a non-smoker, defined as not having smoked or used any form of tobacco or non-tobacco products containing nicotine in more than 6 months before Visit 2/Baseline.
7. Subject has a body mass index (BMI) of 19 to 32 kg/m2 inclusive and body weight not less than 50 kg at Visit 1/Screening.
8. Subject agrees to continue his other general skin care products and regimen for at least 2 weeks prior to Visit 2/Baseline, and through the entire study.
9. Subjects who are sexually active with a female partner and are not surgically sterile (vasectomy performed at least 6 months prior to treatment) must agree to refrain from sperm donation for at least 90 days after application of their last dose of IP and inform their non-pregnant female sexual partner to use a highly effective method of birth control as described in the informed consent form. Note: Male subject must verbally confirm that any female partner(s) must be non-pregnant at Visit 1/Screening and Visit 2/Baseline or at the visit when a subject identifies a new sexual partner.

Exclusion Criteria:

A subject is ineligible to enter the study if he/she meets 1 or more of the following criteria:

1. Subject has any dermatological disorders of the skin within 20 cm of the Treatment Areas with the possibility of interfering with the application of the IP or examination method, such as fungal or bacterial infections, psoriasis, eczema, folliculitis, notable scarring (linear scar > 2.5 cm, etc.), or skin atrophy at Visit 2/Baseline.
2. Subject has any skin pathology or condition that, in the investigator's opinion, could interfere with the evaluation of the IP or requires use of interfering topical, systemic, or surgical therapy at Visit 2/Baseline.
3. Subject has any visible inflammatory skin disease, injury, or condition of their skin that could compromise subject safety and/or interfere with the evaluation of local or systemic assessments performed during the study.
4. Subject has a known or suspected malignancy at Visit 2/Baseline excluding basal cell skin cancer unless it is associated with the Treatment Areas per Exclusion Criterion #1.
5. Subject has a positive blood screen for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C antibody.
6. Subject has any condition, which, in the investigator's opinion, would make it unsafe for the subject to participate in this study, including clinically significant abnormal laboratory, or 12-lead electrocardiogram (ECG) findings during the screening period or Visit 2/Baseline prior to dosing of the IP.
7. Subject has a hospital admission or major surgery within 30 days prior to Visit 2/ Baseline or planned for during the study.
8. Subject is currently enrolled in an investigational drug, biologic, or device study.
9. Subject has used an investigational drug, investigational biologic, or investigational device treatment within 30 days or 5 half-lives, whichever is longer, prior to Visit 2/Baseline.
10. Subject has a history of prescription drug abuse, or illicit drug use within 6 months prior to Visit 1/Screening.
11. Subject has a history of alcohol abuse according to medical history within 6 months prior to Visit 1/Screening.
12. Subject has a positive screen for alcohol or drugs of abuse at Visit 1/Screening or Visit 2/Baseline.
13. Subject has a donation or blood collection of more than 1 unit (approximately 450 mL) of blood (or blood products) or acute loss of blood during the 90 days prior to Visit 2/Baseline.
14. Subject has used systemic prescription medications, herbal (including St John's Wort, herbal teas and garlic extracts) supplements within 14 days prior to dosing at Visit 2/Baseline.
15. Subject has used systemic over-the-counter (OTC) medications or vitamins within 7 days prior to dosing at Visit 2/Baseline. (Note: Use of acetaminophen at < 3g/day is permitted until 24 hours prior to dosing at Visit 2/Baseline).
16. Subject has used topical cosmetic (excluding bland moisturizers), herbal, OTC or prescription products within the designated Treatment Areas 1 day prior to dosing at Visit 2/Baseline.
17. Subject received a live or live attenuated vaccine within 4 weeks of dosing at Visit 2/Baseline.
18. Subject has signs or symptoms consistent with COVID-19 at Visit 1/Screening or Visit 2/Baseline or has been diagnosed with COVID-19 within 4 weeks of Visit 1/Screening.
19. Subject is unable to communicate or cooperate with the investigator due to language problems, poor mental development, or impaired cerebral function.
20. Subject has previously been treated with the IP.
21. Subject has a history of sensitivity to any of the ingredients in the IP.
22. Subject has ongoing or recent history of any other uncontrolled and/or clinically significant systemic disease or condition which, in the investigator's opinion, should exclude participation in the study.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 58 (Actual)
Dates: Start 2023-02-08 (Actual); Primary Completion 2023-08-18 (Actual); Study Completion 2023-10-13 (Actual)

PRIMARY OUTCOMES:
Incidence (severity and causality) of any local and systemic AEs | 42 days
  Collection of adverse events
Number of subjects with presence (and severity) of local skin reactions (LSRs) | 42 days
  Collection of LSRs
Changes from baseline in vital signs-SAD group | 3 days
  Collection of vital signs on day 1 (pre-dose and 6 hrs post-dose) and day 3
Changes from baseline in vital signs-MAD group | 28 days
  Collection of vital signs on day 1, day 7, and day 28
Changes from baseline in laboratory test results-SAD group | 3 days
  Collection of safety labs on day 1, day 2 and day 3
Changes from baseline in laboratory test results-MAD group | 28 days
  Collection of safety labs on day 1, day 7, day 14, and day 28
Changes from baseline in ECG readings-SAD group | 3 days
  Collection of ECGs on day 1 (pre-dose and 6 hrs post-dose) and day 3
Changes from baseline in ECG readings-MAD group | 28 days
  Collection of ECGs on day 1, day 7, and day 28 (pre-dose and 6 hrs post-dose)

SECONDARY OUTCOMES:
Plasma concentrations of TDM-180935 | 29 days
  Plasma concentrations of TDM-180935

CONTACTS AND LOCATIONS:
Overall Officials: Daniel J. Piacquadio, M.D., Study Director — Therapeutics Incorporated
Locations (1):
- TKL Research, Inc., Fair Lawn, New Jersey, United States